CLINICAL TRIAL: NCT00067951
Title: An Open-label Trial to Evaluate the Safety and Efficacy of Fixed Dose Rosiglitazone/Metformin Combination Therapy in Poorly-controlled Subjects With Type 2 Diabetes Mellitus
Brief Title: A Study To Evaluate The Safety And Efficacy Of An Investigational Diabetes Drug In Poorly Controlled Type II Diabetics
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 712753/004
Record Dates: First submitted 2003-09-03; First posted 2003-09-05 (Estimated); Last update posted 2018-03-21 (Actual); Status verified 2018-03

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Hyperglycemia; HbA1c; Hemoglobin A1c; Type 2 diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hyperglycemia | interventions — rosiglitazone-metformin combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: rosiglitazone/metformin

SUMMARY:
The purpose of this research study is to determine if a new investigational diabetes drug is safe and effective in treating people who have Type II diabetes mellitus with very high HbA1c or FPG (fasting plasma glucose) levels. The HbA1c test, also called the hemoglobin A1c test or glycated hemoglobin test, is a measurement of the average amount of sugar in the blood over the last 2 to 3 months. FPG is a test that measures the amount of sugar in the blood after an 8 hour fast.

ELIGIBILITY:
Inclusion Criteria:

* Laboratory result for HbA1c >11% or FPG >270mg/dL
* Clinical diagnosis of Type II diabetes
* Prior treatment with diet and/or exercise alone, or less than 15 days of prior treatment with an oral anti-diabetic medication or insulin.

Exclusion Criteria:

* Women who are pregnant

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2003-10-17; Primary Completion 2004-11-01 (Actual); Study Completion 2004-11-30 (Actual)

PRIMARY OUTCOMES:
Hemoglobin A1c (HbA1c) reduction after 24 weeks of treatment.

SECONDARY OUTCOMES:
Change in FPG, insulin,C-peptide, insulin sensitivity,beta cell function, free fatty acids, lipids. Change in weight, vital signs, clinical laboratory tests, and adverse experiences.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (85):
- United States (44):
  - GSK Investigational Site, Anniston, Alabama
  - GSK Investigational Site, Chandler, Arizona
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Encinitas, California
  - GSK Investigational Site, Fullerton, California
  - GSK Investigational Site, Los Banos, California
  - GSK Investigational Site, Mission Viejo, California
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Melbourne, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Saint Cloud, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Fayetteville, Georgia
  - GSK Investigational Site, Woodstock, Georgia
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Evansville, Indiana
  - GSK Investigational Site, Newburgh, Indiana
  - GSK Investigational Site, Slidell, Louisiana
  - GSK Investigational Site, Jackson, Mississippi
  - GSK Investigational Site, Chesterfield, Missouri
  - GSK Investigational Site, Kansas City, Missouri
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Kingston, New York
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Rochester, New York
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Mogadore, Ohio
  - GSK Investigational Site, Downingtown, Pennsylvania
  - GSK Investigational Site, Warminster, Pennsylvania
  - GSK Investigational Site, West Chester, Pennsylvania
  - GSK Investigational Site, Johnson City, Tennessee
  - GSK Investigational Site, Arlington, Texas
  - GSK Investigational Site, Beaumont, Texas
  - GSK Investigational Site, Bryan, Texas
  - GSK Investigational Site, Corpus Christi, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Midland, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Seattle, Washington
  - GSK Investigational Site, Spokane, Washington
  - GSK Investigational Site, Wenatchee, Washington
- Australia (9):
  - GSK Investigational Site, Camperdown, New South Wales
  - GSK Investigational Site, St Leonards, New South Wales
  - GSK Investigational Site, Wollongong, New South Wales
  - GSK Investigational Site, Kippa-Ring, Queensland
  - GSK Investigational Site, Woolloongabba, Queensland
  - GSK Investigational Site, North Adelaide, South Australia
  - GSK Investigational Site, Caulfield, Victoria
  - GSK Investigational Site, Fremantle, Western Australia
  - GSK Investigational Site, Perth, Western Australia
- Canada (25):
  - GSK Investigational Site, Calgary, Alberta
  - GSK Investigational Site, Coquitlam, British Columbia
  - GSK Investigational Site, Langley, British Columbia
  - GSK Investigational Site, Moncton, New Brunswick
  - GSK Investigational Site, Halifax, Nova Scotia
  - GSK Investigational Site, Brampton, Ontario
  - GSK Investigational Site, Burlington, Ontario
  - GSK Investigational Site, Courtice, Ontario
  - GSK Investigational Site, Kitchener, Ontario
  - GSK Investigational Site, North Bay, Ontario
  - GSK Investigational Site, Oshawa, Ontario
  - GSK Investigational Site, Peterborough, Ontario
  - GSK Investigational Site, Renfrew, Ontario
  - GSK Investigational Site, Stoney Creek, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Laval, Quebec
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Plessisville, Quebec
  - GSK Investigational Site, Pointe-Claire, Quebec
  - GSK Investigational Site, Saint Insidore de Dorchester, Quebec
  - GSK Investigational Site, Saint-Marc-des-Carrieres, Quebec
  - GSK Investigational Site, Sainte Jerome, Quebec
  - GSK Investigational Site, Sherbrooke, Quebec
  - GSK Investigational Site, Regina, Saskatchewan
  - GSK Investigational Site, Saskatoon, Saskatchewan
- New Zealand (4):
  - GSK Investigational Site, Auckland
  - GSK Investigational Site, Christchurch
  - GSK Investigational Site, Rotorua
  - GSK Investigational Site, Wellington
- South Korea (3):
  - GSK Investigational Site, Pusan
  - GSK Investigational Site, Seoul
  - GSK Investigational Site, Uijeongbu-si

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: 712753/004 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 712753/004 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 712753/004 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 712753/004 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 712753/004 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 712753/004 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 712753/004 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register